CLINICAL TRIAL: NCT00815087
Title: Efficacy of Functional Electrical Stimulation in Dysphagia of Nasopharyngeal Cancer Post Radiotherapy
Brief Title: Functional Electrical Stimulation in Irradiated Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200804032R
Record Dates: First submitted 2008-12-25; First posted 2008-12-29 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Dysphagia
Keywords: Nasopharyngeal carcinoma; functional electrical stimulation
MeSH Terms: conditions — Deglutition Disorders; Nasopharyngeal Carcinoma | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional Electrical Stimulation (FES) (Experimental): Functional electrical stimulation: Experimental
  Interventions: Device: Functional electrical stimulation
- Home Rehabilitation Program (HRP) (Active Comparator): Exercise home program
  Interventions: Behavioral: Exercise home program

INTERVENTIONS:
Device: Functional electrical stimulation — 15 sessions of VitalStim® therapy, 60 minutes per session
  Other Names: VitalStim®
  Arms: Functional Electrical Stimulation (FES)
Behavioral: Exercise home program — Daily exercise training
  Other Names: Range of motion exercises, resistence exercises, etc...
  Arms: Home Rehabilitation Program (HRP)

SUMMARY:
The purpose of this study is to determine whether functional electrical stimulation is effective in the treatment of dysphagia due to nasopharyngeal cancer post radiotherapy

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) patients usually underwent radiotherapy (RT) or chemoradiotherapy(CRT). There were some complications caused by RT, like dysphagia.

In recent studies, functional electrical stimulation (FES) was be used in neurologically dysphagia patients, and there were some positive effects with these studies. Hence, we decided applied FES to these NPC patients with dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Primary nasopharyngeal carcinoma
* Post radiation therapy
* Mild to severe dysphagia
* Never underwent swallowing therapy

Exclusion Criteria:

* Recurrent cancer
* Neurological or degenerate disease
* Total or partial laryngectomy
* Epilepsy
* With cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyng-Guey Wang, MD, Principal Investigator — Department of Physicale Medicine and Rehabilitation, National Taiwan University Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty subjects were referral from department of oncology & physical Medicine and Rehabilitation, National Taiwan University Hospital, Taipei, Taiwan. The study was approved by the Ethics Committee of the National Taiwan University Hospital. All participants gave their informed consent.
Pre-assignment Details: They were assigned into the FES group and home rehabilitation program (HRP) group by the method of sex stratified randomization, and were matched by Dysphagia Outcome and Severity Scale (DOSS) score within 1 unit in order to compare two groups under the same sex proportion and similar DOSS score pairs.
Groups:
- Functional Electrical Stimulation (FES): Functional electrical stimulation: Experimental
  Functional electrical stimulation : 15 sessions of VitalStim® therapy, 60 minutes per session
- Home Rehabilitation Program (HRP): Exercise home program
  Exercise home program : Daily exercise training
Period: Overall Study
Arm/Group | Functional Electrical Stimulation (FES) | Home Rehabilitation Program (HRP)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We decided to make the cut point when the numbers of 2 groups are equal.
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Electrical Stimulation (FES) | Home Rehabilitation Program (HRP) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (7.4) | 56.1 (11.8) | 54.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Taiwan | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline and Cut Point VFSS in Velocity of Displacement of Hyoid Bone at 1 to 3 Months
Description: A parameter of the VFSS assessment was velocity of displacement of hyoid bone on 5mL thin barium sulfate bolus, which was defined as the displacement divided by the duration. The outcome measure time frame was based on VFSS assessment with the range between one to three months due to subjects received 1 to 3 times per week. We will provide the mean time frame, which is 2 months.
Time Frame: Averaged 2 months
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Functional Electrical Stimulation (FES) | Home Rehabilitation Program (HRP)
Number analyzed (Participants) | 10 | 10
cm/s | 0.8 (0.5) | -0.4 (0.8)

2. Secondary Outcome: Questionnaire of Life Quality
Time Frame: 1 to 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The data were collected from cut point VFSS to 1 year.
Description: Not any patient reported serious adverse event.
Arm/Group | Functional Electrical Stimulation (FES) | Home Rehabilitation Program (HRP)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Lack of information about muscle fibrosis, no control group. and the results from the small amount of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes